CLINICAL TRIAL: NCT02490111
Title: Efficacy and Safety of DWJ1319 in the Prevention of Gallstone Formation After Gastrectomy in Patient With Gastric Cancer: A Multicenter, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Clinical Trials for the Prevention of Gallstone Formation After Gastrectomy in Patient With Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DW_UDCA005
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- DWJ1319 300 mg BID (Experimental): DWJ1319 300 mg, orally, twice daily (BID) for up to 12 months
  Interventions: Drug: DWJ1319
- DWJ1319 300 mg QD (Experimental): DWJ1319 300 mg, orally, once daily (QD), and DWJ1319 placebo-matching capsules, orally, once daily for up to 12 months
  Interventions: Drug: DWJ1319; Drug: Placebo
- Placebo (Placebo Comparator): Placebo, orally, twice daily (BID) for up to 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWJ1319
  Arms: DWJ1319 300 mg BID; DWJ1319 300 mg QD
Drug: Placebo
  Arms: DWJ1319 300 mg QD; Placebo

SUMMARY:
This study evaluates the efficacy and safety of DWJ1319 in the prevention of gallstone formation after gastrectomy in patient with gastric cancer. Two-thirds of the participants will receive DWJ1319, while the other will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 19 years of age
* Patient who undergoes gastrectomy (total, distal or proximal gastrectomy)
* D1+ or D2 lymph node dissection
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* Written informed consent

Exclusion Criteria:

* Patients with cholangitis, cholecystitis, non-functional gall bladder, or biliary obstruction
* Presence of gallstones on ultrasonography and/or CT
* History of previous cholecystectomy
* Patients undergoing pylorus-preserving gastrectomy
* Pregnant or lactating women and fertile women who is not using proper contraceptive method
* Patients with history of drug or alcohol abuse within 5 years ago

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patient developing gallstone at 12 month after gastrectomy | 12 months

SECONDARY OUTCOMES:
Proportion of patient developing gallstone at 3, 6 and 9 month after gastrectomy | 3, 6 and 9 months
Time to gallstone formation | 12 months

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul Natioanl University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Pusan National University Yangsan Hospital, Yangsan, Kyeongsangnamdo
  - Kyungpook National university Chilgok Hospital, Daegu
  - Chungnam National university hospital, Daejeon
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Lee SH, Jang DK, Yoo MW, Hwang SH, Ryu SY, Kwon OK, Hur H, Man Yoon H, Eom BW, Ahn HS, Son T, Song KY, Lee HH, Choi MG, An JY, Lee SI, Lee KH, Ahn S, Park YS, Park DJ; Efficacy and Safety of DWJ1319 in the Prevention of Gallstone Formation after Gastrectomy in Patient with Gastric Cancer: A Multicenter, Randomized, Double-blind, Placebo-controlled Study (PEGASUS-D) Group. Efficacy and Safety of Ursodeoxycholic Acid for the Prevention of Gallstone Formation After Gastrectomy in Patients With Gastric Cancer: The PEGASUS-D Randomized Clinical Trial. JAMA Surg. 2020 Aug 1;155(8):703-711. doi: 10.1001/jamasurg.2020.1501. PMID 32584935